CLINICAL TRIAL: NCT03133793
Title: Reducing Symptom Burden in Patients With Heart Failure With Preserved Ejection Fraction Using Ubiquinol and/or D-ribose
Brief Title: CoQ10 and D-ribose in Patients With Diastolic Heart Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00140741; 5R01AG054486-02 (NIH)
Record Dates: First submitted 2017-04-25; First posted 2017-04-28 (Actual); Results first posted 2022-03-03 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Heart Failure, Diastolic
Keywords: heart failure with preserved ejection fraction
MeSH Terms: conditions — Heart Failure, Diastolic | interventions — coenzyme Q10

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo Only (Placebo Comparator): Participants in this group will receive placebo pills and placebo powder.
  Interventions: Other: Placebo pills; Other: Placebo powder
- CoQ10 Only (Active Comparator): Participants in this group will receive CoQ10 pills and placebo powder
  Interventions: Drug: CoQ10; Other: Placebo powder
- D-ribose Only (Active Comparator): Participants in this group will receive placebo pills and D-ribose oral powder.
  Interventions: Drug: D-Ribose Oral Powder; Other: Placebo pills
- CoQ10 + D-ribose (Experimental): Participants in this group will receive CoQ10 pills and D-ribose oral powder.
  Interventions: Drug: CoQ10; Drug: D-Ribose Oral Powder

INTERVENTIONS:
Drug: CoQ10 — Participants will take 300 mg capsules two times daily, 1 taken in the morning and 1 taken in the evening, for up to 12 weeks.
  Arms: CoQ10 + D-ribose; CoQ10 Only
Drug: D-Ribose Oral Powder — Participants will mix 15 grams D-Ribose powder, mixed with non-carbonated liquid, one time per day for up to 12 weeks.
  Arms: CoQ10 + D-ribose; D-ribose Only
Other: Placebo pills — Participants will take matched placebo pills that are 300 mg capsules, two times daily, 1 taken in the morning and 1 taken in the evening, for up to 12 weeks.
  Arms: D-ribose Only; Placebo Only
Other: Placebo powder — Participants will mix 15 grams placebo powder, mixed with non-carbonated liquid, one time per day for up to 12 weeks.
  Arms: CoQ10 Only; Placebo Only

SUMMARY:
The purpose of this study is to compare the clinical benefits of CoQ10 and D-ribose taken by patients who have diastolic heart failure, or heart failure with preserved ejection fraction (HFpEF).

DETAILED DESCRIPTION:
This study used a novel design to compare ubiquinol and/or D-ribose as supplemental treatments for HFpEF using a biobehavioral model. This was a randomized, double-blind, controlled trial with a total sample size of (N) = 216 All participants received usual care for HFpEF. Efforts were made to recruit 50% females which is the actual proportion of HFpEF patients in Kansas City area. There were 63 subjects that did not make the 7 day enrollment which dropped our participants to 153.

Participants in this study were randomized into 4 study groups (total n = 153):

N1 = 39 subjects: Control, receive no ubiquinol and no D-ribose; placebo capsules & powder per day.

N2 = 39 subjects: Ubiquinol group, receive 600 mg of ubiquinol/day, D-ribose placebo powder per day.

N3 = 37 subjects: D-ribose group, receive 15 g of D-ribose/day, placebo capsules for ubiquinol per day.

N4 = 38 subjects: Ubiquinol + D-ribose group, receive 600 mg ubiquinol and 15 g D-ribose per day.

The enrolled patients were randomized into four groups to receive ubiquinol (600 mg daily), D-ribose (15 g daily), ubiquinol plus D-ribose, or placebo for a period lasting 12 weeks. Both the ubiquinol and the D-ribose supplements used in the study had a certificate of analysis from the manufacturer. The Project Manager reviewed the electronic health records at the University of Kansas Health System (TUKHS) to identify subjects that met the study criteria and were approached to study inclusion. Once the subject signed the informed consent and successfully completed the 7-day run-in, they were randomly assigned to one of the four groups using a list created by a computer-based random number generator. All supplements and the placebo were indistinguishable in packaging and were distributed by the Project Manager or Research Associate independent of the PI so that the allocation of subjects to a treatment or placebo group were concealed from both subjects and key research personnel.

All subjects arrived at the Clinical and Translational Science Unit (CTSU) and escorted to a private exam room. They completed the demographic form at baseline. The KCCQ and Vigor scale from the Profile of Mood States (POMS) were completed in CTSU visits at baseline, and 12 weeks along with the subject's blood pressure, heart rate, height, and weight. The patient was given privacy and asked to remove clothing above the waist. A disposable gown was provided, and the patient laid supine on the bed while an echocardiogram was completed. Approximately, 1 ml of blood was drawn to measure lactate. adenosine triphosphate (ATP), and B-type natriuretic peptide (BNP). The blood samples were measured with point-of-contact instruments within 5 minutes at the CTSU. After the echocardiogram, questionnaires, BNP, and ATP measurements, the subjects completed the six-minute walk test (6MWT) with the Borg scale. The entire data collection period was approximately 2 hours for each subject's visit to the CTSU. Follow-up calls occurred at 3, 6, and 9 weeks during the trial.

Various cardiovascular risk factors were recorded such as tobacco usage, diabetes mellitus, hypercholesterolemia, hypertension, and family history of cardiovascular disease. Smoking status was recorded as either smoker or non-smoker. Diabetes mellitus was also determined by a history of the disease or use of medication for diabetes. Hypercholesterolemia was defined as a fasting total serum cholesterol level ≥ 4.9 mmol/l or use of medication. Hypertension was defined as either systolic or diastolic blood pressure ≥ 140/90 mmHg or use of hypertensive medications.

Aims and Hypotheses.

There were 2 aims and 6 hypotheses:

AIM #1: To determine the effects of oral ubiquinol, D-ribose, or a combination of the two administered during 12 weeks on symptoms accompanying low bioenergetics in patients with HFpEF.

Hypothesis #1. Ubiquinol (600 mg daily), D-ribose (15 g daily), or a combination of the two will enhance the health status of patients with HFpEF as measured by the Kansas City Cardiomyopathy Questionnaire (KCCQ).

Primary outcomes of the study were patient-centered; thus the measurement of health status was a priority. Bioenergetics has both biological and behavioral components. The biological component (i.e., improved heart function) and its measurement was discussed in Aim #2.

Investigators assessed patients' perceptions of their symptoms using the KCCQ, a self-administered questionnaire that measures patients' perceptions of five domains of their health status relevant to HFpEF. These domains are: (1) physical limitations, (2) symptoms, (3) self-efficacy, (4) quality of life, and (5) social interference. The KCCQ consists of 24 items to which patients respond on a scale indicating limitations due to HF. For example, for activities such as dressing, doing yard work, or climbing a flight of stairs, patients were asked to check a response that indicates the degree to which HF has limited their ability: "Extremely Limited," "Quite a bit Limited," "Moderately Limited," "Slightly Limited," "Not at all Limited," or "Limited for other reasons or did not do the activity." Another item is: "Over the past 2 weeks, how many times has shortness of breath limited your ability to do what you wanted?" Response alternatives are: "All of the time," "Several times," "At least once a day," "3 or more times per week but not every day," "1-2 times per week," "Less than once a week," and "Never over the past 2 weeks." The KCCQ takes only 4 to 6 minutes to complete and has been used in more than a hundred studies. It has excellent psychometric properties and clinical usefulness including: (1) high test-retest reliability; (2) high internal consistency within each area (e.g., Cronbach's alpha ranged from 0.78 to 0.90); (3) patients' scores concerning their health status correlate well with objective measurements of their functional capacities; and (4) the scale's sensitivity for detecting clinical changes in HF patients is significantly greater than that of the Minnesota Living with Heart Failure Scale. Investigators used the KCCQ to compare the changes in health status of patients with HFpEF taking ubiquinol, D-ribose, ubiquinol + D-ribose, or placebo.

Hypothesis #2. Ubiquinol (600 mg daily), D-ribose (15 g daily), or a combination of the two will increase the level of vigor in patients with HFpEF as measured by the Vigor subscale of the Profile of Mood States (POMS).

Using the Vigor subscale from the POMS questionnaire, patients rated themselves on eight adjectives (lively, active, energetic, cheerful, alert, full of pep, carefree, and vigorous) on a five-point scale (0 = not at all, 1 = a little, 2 = moderately, 3 = quite a bit, and 4 = extremely). The Vigor scale has very high internal consistency (Cronbach's alpha = 0.90), and it takes only 1 minute to complete. In many studies it has been found to be effective for assessing vigor changes associated with exercise. The KCCQ and POMS Vigor scale were administered to patients after they have been sitting quietly for 10 minutes at the beginning of each visit (baseline, 12 weeks). The total time for patients to complete both questionnaires was 5 to10 minutes.

AIM #2: To determine the effects of oral ubiquinol, D-ribose, or a combination of the two over 12 weeks on biological measures in patients with HFpEF.

Hypothesis #3. Ubiquinol (600 mg daily), D-ribose (15 g daily), or a combination of the two will improve left ventricular diastolic function measured by advanced echocardiographic imaging in patients with HFpEF.

Two-dimensional Doppler echocardiography was used for myocardial imaging to assess cardiac function in patients with HFpEF. In this study, a echocardiography technician performed the echocardiograms during each visit (baseline and 12 weeks). Dr. Hiebert (cardiologists) determine ejection fraction (EF) and the ratio of mitral peak velocity of early filling (E) to early diastolic mitral annular velocity (eꞌ) (E/eꞌ ratio) (SV, EDV, EF) from the echocardiogram.

Hypothesis #4. Ubiquinol (600 mg daily), D-ribose (15 g daily), or a combination of the two will increase the distance that patients with HFpEF can walk in 6 minutes.

Investigators examined the effects of ubiquinol and/or D-ribose on the 6MWT at baseline and 12 weeks. Participants were asked to wear appropriate clothes and shoes and walk the longest distance possible in 6 minutes. Prior to exercising, there was a 10-minute rest period during which heart rate and blood pressure were recorded. Subjects walked indoors on a flat, straight 30-meter path marked every 3 meters, and they were informed that they could slow down or stop at any time. A one-lap demonstration was completed before the test began. The distance walked was recorded. Following the 6MWT, a 0.5 ml blood sample was obtained for lactate measurement. Lactate provides a measure of the oxygen debt occurring during exercise and correlates directly with reported dyspnea and fatigue. The patient also recorded perceived dyspnea and fatigue at baseline and at the end of each walk by using the Borg scale, where 0 = nothing at all, 5 = severe, and 10 = very severe.

Hypothesis #5. Ubiquinol (600 mg daily), D-ribose (15 g daily), or a combination of the two will decrease venous blood B-type natriuretic peptide (BNP) levels in patients with HFpEF.

BNP concentration was measured using a portable i-STAT handheld analyzer. A blood sample (20 μl) was obtained from a finger stick after the subjects have completed the questionnaires at baseline and 12 weeks. Investigators measured BNP concentration at each visit.

Hypothesis #6. Ubiquinol (600 mg daily), D-ribose (15 g daily), or a combination of the two will decrease the lactate/ATP ratio in patients with HFpEF.

0.1 ml blood sample obtained by finger stick was used for ATP measurements (AquaSnap Total system) after the subject had completed the questionnaires and echocardiograms. Lactate concentration was measured after the 6MWT with a portable i-STAT handheld instrument and requires 0.5 ml blood.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with HFpEF within a 6-month period
* New York Heart Association (NYHA) Classification II-III HF
* Have left ventricular ejection fraction (EF) ≥ 50% documented by an echocardiogram
* Have a telephone or reliable phone contact
* Have their own means of transportation to the study site

Exclusion Criteria:

* Acute coronary syndrome in the past 12 weeks
* Significant valvular heart disease
* Severe cardiac fibrosis (galectin-3 level > 26 ng/ml)
* Constrictive pericardium
* Pulmonary fibrosis
* Congenital heart disease
* Hypertrophic or infiltrative cardiomyopathy
* Heart transplant
* Left ventricular assist device
* Heart failure (HF) associated hospital admission or emergency room visit within past 30 days
* Recent percutaneous coronary intervention
* Significant renal and/or hepatic dysfunction
* Severe cognitive impairment
* Consumption of any CoQ10 (ubiquinol) or D-ribose supplements

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2021-03-12 (Actual); Study Completion 2021-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet Pierce, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No
None at this time.

REFERENCES:
- [Derived] Pierce JD, Shen Q, Mahoney DE, Rahman F, Krueger KJ, Diaz FJ, Clark L, Smith C, Vacek J, Hiebert JB. Effects of Ubiquinol and/or D-ribose in Patients With Heart Failure With Preserved Ejection Fraction. Am J Cardiol. 2022 Aug 1;176:79-88. doi: 10.1016/j.amjcard.2022.04.031. Epub 2022 May 27. PMID 35644694
- [Derived] Pierce JD, Mahoney DE, Hiebert JB, Thimmesch AR, Diaz FJ, Smith C, Shen Q, Mudaranthakam DP, Clancy RL. Study protocol, randomized controlled trial: reducing symptom burden in patients with heart failure with preserved ejection fraction using ubiquinol and/or D-ribose. BMC Cardiovasc Disord. 2018 Apr 2;18(1):57. doi: 10.1186/s12872-018-0796-2. PMID 29606104

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment started for this clinical trial February 5, 2018 and recruitment occurred at The University of Kansas Hospital in the cardiology and heart failure clinics.
Pre-assignment Details: Trial included a 7 day run-in period where the participant was asked to take placebo capsules and powder. They had to consume 80% of both placebo items to be randomized into the study. There were many subjects who signed the consent form and started on the run-in period but never returned for data collection (n=63).
Groups:
- Placebo Only: Participants in this group received placebo pills and placebo powder.
  Placebo pills: Participants took matched placebo pills that were 300 mg capsules, two times daily, 1 taken in the morning and 1 taken in the evening, for up to 12 weeks.
  Placebo powder: Participants mixed 15 grams placebo powder, mixed with non-carbonated liquid, one time per day for up to 12 weeks.
- CoQ10 (Ubiquinol) Only: Participants in this group received CoQ10 (ubiquinol) capsules and placebo powder
  CoQ10 (Ubiquinol): Participants took 300 mg capsules two times daily, 1 taken in the morning and 1 taken in the evening, for up to 12 weeks.
  Placebo powder: Participants mixed 15 grams placebo powder, mixed with non-carbonated liquid, one time per day for up to 12 weeks.
- D-ribose Only: Participants in this group received placebo pills and D-ribose oral powder.
  D-Ribose Oral Powder: Participants mixed 15 grams D-Ribose powder, mixed with non-carbonated liquid, one time per day for up to 12 weeks.
  Placebo pills: Participants took matched placebo pills that are 300 mg capsules, two times daily, 1 taken in the morning and 1 taken in the evening, for up to 12 weeks.
- CoQ10 (Ubiquinol) + D-ribose: Participants in this group received CoQ10 (ubiquinol) capsules and D-ribose oral powder.
  CoQ10 (Ubiquinol): Participants took 300 mg capsules two times daily, 1 taken in the morning and 1 taken in the evening, for up to 12 weeks.
  D-Ribose Oral Powder: Participants mixed 15 grams D-Ribose powder, mixed with non-carbonated liquid, one time per day for up to 12 weeks.
Period: Overall Study
Arm/Group | Placebo Only | CoQ10 (Ubiquinol) Only | D-ribose Only | CoQ10 (Ubiquinol) + D-ribose
Started | 39 | 39 | 37 | 38
Completed | 38 | 35 | 33 | 33
Not Completed | 1 | 4 | 4 | 5
Not completed — Withdrawal by Subject | 0 | 4 | 2 | 4
Not completed — Lost to Follow-up | 1 | 0 | 2 | 0
Not completed — Death | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Only | CoQ10 Only | D-ribose Only | CoQ10 + D-ribose | Total
Number analyzed (Participants) | 39 | 39 | 37 | 38 | 153
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 12 | 14 | 12 | 49
  >=65 years | 28 | 27 | 23 | 26 | 104
Age, Continuous [Median (Standard Deviation); unit: years] | 69.0 (9.3) | 67.0 (10.6) | 72.0 (10.6) | 69.5 (9.4) | 69 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 21 | 22 | 20 | 86
  Male | 16 | 18 | 15 | 18 | 67
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity : Hispanic or Latino | 1 | 3 | 1 | 4 | 9
  Ethnicity : Non-Hispanic | 37 | 36 | 36 | 34 | 143
  Ethnicity : Unknown | 1 | 0 | 0 | 0 | 1
  Race : African American | 7 | 7 | 6 | 6 | 26
  Race: American Indian or Alaska Native | 0 | 0 | 1 | 2 | 3
  Race: Asian | 0 | 0 | 0 | 1 | 1
  Not Reported | 0 | 0 | 0 | 1 | 1
  Other | 0 | 2 | 1 | 1 | 4
  White | 32 | 30 | 29 | 27 | 118
Region of Enrollment [Number; unit: participants]
  United States | 39 | 39 | 37 | 38 | 153
Kansas City Cardiomyopathy Questionnaire [Mean (Standard Deviation); unit: units on a scale] — The KCCQ has a 2-week recall period of heart failure symptoms with 23 items that map to 7 domains: symptom frequency; symptom burden; symptom stability; physical limitations; social limitations; quality of life; and self-efficacy. The total symptom score is combined with the physical limitations for a clinical summary score. All scores are represented on a 0-to-100-point scale. Lower scores represent more severe symptoms and/or limitations and scores of 100 indicate no symptoms, no limitations, excellent quality of life and better health status.
  units on a scale | 48.52 (24.23) | 51.88 (23.17) | 44.05 (19.11) | 45.63 (21.6) | 47.52 (22.03)
Vigor Scale [Mean (Standard Deviation); unit: units on a scale] — The Vigor subscale of the Profile of Mood States (POMS). questionnaire is where the patients rate themselves on eight adjectives (lively, active, energetic, cheerful, alert, full of pep, carefree, and vigorous) on a five-point scale (0 = not at all, 1 = a little, 2 = moderately, 3 = quite a bit, and 4 = extremely). Scores for the subscale range from 0-32, in which higher scores reflect more vigor and lower scores reflect less vigor. The Vigor scale has very high internal consistency (Cronbach's alpha = 0.90), and it takes only 1-2 minute to complete.
  units on a scale | 13.79 (5.7) | 13 (5.49) | 13.94 (7.11) | 12.21 (5.57) | 13.24 (5.97)
Ejection Fraction (EF) [Mean (Standard Deviation); unit: percentage of ejection fraction] — Ejection fraction (EF) is a measurement expressed as a percentage of how much blood the left ventricle pumps out with each contraction. Population: With some patients that were obese, we could obtain an ejection fraction but not an septal E/e' value.
  percentage of ejection fraction
    number analyzed (Participants) | 37 | 33 | 31 | 32 | 133
    (all) | 51.04 (7.43) | 51.89 (5.68) | 50.79 (4.38) | 51.28 (4.76) | 51.25 (5.56)
6-minute walking test (6MWT) [Mean (Standard Deviation); unit: meters] — The six minute walking test (6MWT) is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity. Population: Some participants were unable to walk that day. They either did not feel well or forgot to wear proper shoes so they did not want to walk.
  meters
    number analyzed (Participants) | 38 | 34 | 33 | 33 | 138
    (all) | 247.87 (150.96) | 322.69 (124.18) | 265.58 (135.96) | 237.85 (131.05) | 268.49 (135.54)
B-type natriuretic peptide (BNP) level [Mean (Standard Deviation); unit: pg/mL] — Population: Some of the participants we were unable to obtain a blood sample or they refused.
  pg/mL
    number analyzed (Participants) | 38 | 35 | 33 | 32 | 138
    (all) | 232 (388.28) | 182.51 (211.23) | 152.48 (141.52) | 157.09 (155.27) | 181.02 (224.08)
lactate [Mean (Standard Deviation); unit: mmol/L] — Population: During the participant visit we either had instrument error or the patient did not want us to stick them again.
  mmol/L
    number analyzed (Participants) | 38 | 35 | 33 | 31 | 137
    (all) | 2.45 (1.13) | 2.58 (1.04) | 2.34 (1.12) | 2.72 (1.59) | 2.52 (1.22)
Septal E/e' [Mean (Standard Deviation); unit: ratio] — Early diastolic mitral annulus velocity (e') estimated by tissue Doppler and the ratio of the transmitral early peak velocity (E) by pulsed wave Doppler over e' (E/e') are the two key parameters for grading a diastolic dysfunction as they represent a reliable noninvasive surrogate for left ventricular diastolic pressures. Population: If the patient was obese, it was difficult to obtain a measurement using a 2-D doppler system.
  ratio
    number analyzed (Participants) | 33 | 29 | 28 | 27 | 117
    (all) | 9.41 (5.54) | 9.8 (4.27) | 11.2 (5.97) | 9.35 (4.24) | 9.94 (5.05)
Adenosine Phosphate (ATP) [Mean (Standard Deviation); unit: Relative Light Units (RLU)] — Population: We were unable to obtain blood samples from some subjects due to difficulty obtaining the sample or the patient refusing the test.
  Relative Light Units (RLU)
    number analyzed (Participants) | 38 | 35 | 33 | 33 | 139
    (all) | 3332.87 (844.33) | 3222.63 (1040.44) | 3312.18 (915.98) | 3383.24 (954.03) | 3312.73 (938.695)

OUTCOME MEASURES:

1. Primary Outcome: Change in Health Status of Patients With HFpEF
Description: Patients' perceptions of their symptoms were measured using the Kansas City Cardiomyopathy Questionnaire (KCCQ), a self-administered questionnaire that measures patients' perceptions of five domains of their health status relevant to HFpEF. The KCCQ is a 24 item questionnaire. Scores are transformed to a range of 0-100, in which higher scores reflect better health status. All scores are represented on a 0-to-100-point scale, where lower scores represent more severe symptoms and/or limitations and scores of 100 indicate no symptoms, no limitations, and excellent quality of life.
Time Frame: Change from Baseline to Week 12
Population: A few of the subjects refused to complete the questionnaire or drop out of the study due to COVID-19.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo Only | CoQ10 Only | D-ribose Only | CoQ10 + D-ribose
Number analyzed (Participants) | 37 | 35 | 33 | 33
Scores on a scale | 4.15 (24.04) | 26.56 (18.61) | 29.97 (21.95) | 33 (21.45)

2. Secondary Outcome: Change in Vigor
Description: Change were measured using the the Vigor subscale from the Profile of Mood States (POMS) questionnaire. Patients rated themselves on eight adjectives (lively, active, energetic, cheerful, alert, full of pep, carefree, and vigorous) on a five-point scale (0 = not at all, 1 = a little, 2 = moderately, 3 = quite a bit, and 4 = extremely). Scores for the subscale range from 0-32, in which higher scores of 32 reflected more vigor and a score of 0 reflected no vigor.
Time Frame: Change from Baseline to Week 12
Population: A few of the subjects refused to complete the questionnaire or drop out of the study due to COVID-19.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo Only | CoQ10 Only | D-ribose Only | CoQ10 + D-ribose
Number analyzed (Participants) | 37 | 35 | 33 | 33
Scores on a scale | -0.54 (7.32) | 7.11 (5.1) | 7.3 (6.79) | 7.61 (5.9)

3. Secondary Outcome: Change in Ejection Fraction (EF)
Description: Change was measured using the the ejection fraction using echocardiographic imaging. Ejection fraction (EF) is the percentage of blood volume ejected in each cardiac cycle and is a representation of left ventricular systolic performance.
Time Frame: Change from Baseline to Week 12
Population: Some of the patients were morbidly obese and we were unable to obtain accurate ejection fraction measurements.
Measure: Mean (Standard Deviation); unit: percentage of ejection fraction
Arm/Group | Placebo Only | CoQ10 Only | D-ribose Only | CoQ10 + D-ribose
Number analyzed (Participants) | 36 | 33 | 30 | 30
percentage of ejection fraction | -2.39 (6.96) | 4.69 (7.72) | 5.64 (6.67) | 5.07 (7.14)

4. Secondary Outcome: Change in Septal E/e'
Description: Change was measured using the the Septal E/e' using advanced echocardiographic imaging. Septal E/e' is the early diastolic mitral annulus velocity (e') estimated by tissue Doppler using an echocardiogram and the ratio of the transmitral early peak velocity (E) by pulsed wave Doppler over e' (E/e'). These are the two key parameters for grading a diastolic dysfunction as they represent a reliable noninvasive surrogate for left ventricular diastolic pressures.
Time Frame: Change from Baseline to Week 12
Population: Some of the participants were morbidly obese and we were unable to obtain accurate images.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Placebo Only | CoQ10 (Ubiquinol) Only | D-ribose Only | CoQ10 (Ubiquinol) + D-ribose
Number analyzed (Participants) | 36 | 33 | 30 | 30
ratio | 1.39 (7.74) | -1.27 (4.17) | -0.65 (6.48) | -0.47 (4.40)

5. Secondary Outcome: Change in 6 Minute Walk Test (6MWT)
Description: Change was measured using the 6-minute walking test. The 6-minute walking test (6MWT) is a simple test. Test measures the total distance in meters a person can walk in 6 minutes.
Time Frame: Change from Baseline to Week 12
Population: A few of the subjects were refused to walk due to an injury or drop out of the study due to COVID-19.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Placebo Only | CoQ10 Only | D-ribose Only | CoQ10 + D-ribose
Number analyzed (Participants) | 38 | 34 | 33 | 33
meters | 19.62 (76.27) | 21.21 (36.73) | 29.42 (52.92) | 36.21 (42.28)

6. Secondary Outcome: Change in Venous Blood B-type Natriuretic Peptide (BNP) Levels
Description: Change was measured for brain natriuretic peptide. Brain natriuretic peptide (BNP) levels are objective measures of cardiac function. BNP testing is a useful tool in predicting prognoses in patients with heart failure
Time Frame: Change from Baseline to Week 12
Population: We were unable to obtain blood on a few subjects or they drop out of the study due to COVID-19.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo Only | CoQ10 Only | D-ribose Only | CoQ10 + D-ribose
Number analyzed (Participants) | 38 | 33 | 31 | 29
pg/mL | -18.43 (80.37) | -29.56 (67.43) | -42.94 (72.47) | 29.08 (68.08)

7. Secondary Outcome: Change in Lactate
Description: Change was measured for lactate. Lactate is produced by anaerobic metabolism and may reflect inadequate tissue perfusion in conditions such heart failure with preserved ejection fraction.
Time Frame: Change from Baseline to Week 12
Population: The number analyzed in one or more rows differs because we had either an instrument error or we were unable to obtain an adequate blood sample.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo Only | CoQ10 Only | D-ribose Only | CoQ10 + D-ribose
Number analyzed (Participants) | 38 | 34 | 32 | 31
mmol/L | 0.33 (1.26) | 0 (0.79) | -0.35 (0.7) | -0.24 (0.88)

8. Secondary Outcome: Change in Adenosine Triphosphate (ATP)
Description: All cellular processes require ATP as a primary energy source. The heart requires ATP for the function of membrane transport systems (e.g., Na+/K+-ATPase) as well as for sarcomere contraction and relaxation.
Time Frame: Change from Baseline to Week 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: relative light units (RLU)
Arm/Group | Placebo Only | CoQ10 (Ubiquinol) Only | D-ribose Only | CoQ10 (Ubiquinol) + D-ribose
Number analyzed (Participants) | 38 | 34 | 32 | 31
relative light units (RLU) | -189.08 (828.43) | 1133.5 (997.89) | 907.44 (1006.78) | 686.19 (1018.41)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were assessed every 4 weeks throughout treatment from time of first dose and up to the last day at 12 weeks. AEs were evaluated over treatment which was a maximum duration of 3 cycles (approximately 3 months).
Description: SAEs defined per protocol and all remaining AEs categorized as Other AE without regard to treatment attribution.
Arm/Group | Placebo Only | CoQ10 Only | D-ribose Only | CoQ10 + D-ribose
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/35 | 0/33 | 1/33
Serious Adverse Events (participants affected / at risk) | 8/38 | 10/35 | 5/33 | 7/33
Other Adverse Events (participants affected / at risk) | 2/38 | 1/35 | 1/33 | 2/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Only (N=38) | CoQ10 Only (N=35) | D-ribose Only (N=33) | CoQ10 + D-ribose (N=33)
Heart Failure (Cardiac disorders) | 3 (3) | 2 (2) | 0 (0) | 1 (1)
Chest pain (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Lung Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 3 (3) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pericardial Effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal Colic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Only (N=38) | CoQ10 Only (N=35) | D-ribose Only (N=33) | CoQ10 + D-ribose (N=33)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bullous Dermatitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
One limitation of this clinical trial was the occurrence of the COVID-19 pandemic during data collection. Several of the patients decided not to participate leading to a small number of subjects in the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-22): https://cdn.clinicaltrials.gov/large-docs/93/NCT03133793/Prot_SAP_000.pdf